CLINICAL TRIAL: NCT06776354
Title: Application of Artificial Intelligence in Hypertension Pharmacotherapy Education: A Comparative Study of the GPT System and Traditional Teaching Methods
Brief Title: AI in Hypertension Treatment Education: Comparing GPT and Traditional Methods
Acronym: AIHT-EDU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: zhen wang (Other)
Responsible Party: Sponsor-Investigator, zhen wang, physician-in-charge, The Second Hospital of Anhui Medical University
Organization: The Second Hospital of Anhui Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023jyxm1150; 2023jyxm1150 (Other Grant/Funding Number: 2023 Anhui Province Quality Engineering Project)
Record Dates: First submitted 2024-12-27; First posted 2025-01-15 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-03

CONDITIONS: Medical Education; Hypertension; GPT
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GPT-based training (Experimental): Generative Pre-trained Transformer (GPT)-based training system
  Interventions: Behavioral: GPT-based training
- traditional training (Active Comparator): traditional training method
  Interventions: Behavioral: traditional training

INTERVENTIONS:
Behavioral: GPT-based training — GPT-based training whether could improve the ability of students to develop effective hypertension management plans
  Arms: GPT-based training
Behavioral: traditional training — traditional teaching methods
  Arms: traditional training

SUMMARY:
Educational Trial: GPT-Based Training vs. Traditional Teaching for Hypertension Management

The goal of this educational trial is to determine whether a Generative Pre-trained Transformer (GPT)-based training system is more effective than traditional teaching methods in helping medical students master hypertension management plans. It will also evaluate the educational effectiveness and engagement of the GPT-based system. The main questions it aims to answer are:

Does the GPT-based training improve the ability of students to develop effective hypertension management plans compared to traditional methods? How do students perceive the use of the GPT system in their learning process? Researchers will compare the GPT-based training system to traditional teaching methods to see if the innovative AI approach enhances learning outcomes in medical education.

Participants will:

Engage with either the GPT-based system or traditional teaching materials. Visit the educational facility periodically for assessments and feedback sessions.

Keep a diary of their learning experiences, noting any difficulties or advantages they observe in the training method they are assigned.

ELIGIBILITY:
Inclusion Criteria:

* Graduate or regulatory trainee, currently rotating in cardiology and willing to participate in research.
* Age between 18-30 years old, gender not limited.
* No specialized training experience in hypertension diagnosis and treatment, only possessing basic medical theoretical knowledge.
* Able to accept a 4-week teaching intervention (2 hours of study per week).
* Sign the informed consent form and be aware of the research purpose and process.

Exclusion Criteria:

* Graduate students or trained interns who have received specialized training in hypertension medication treatment.
* Students unable to complete the full course of study (e.g., rotations shorter than four weeks or potential mid-course withdrawal).
* Unable to consistently participate in educational interventions (e.g., conflicts with study schedule).
* Have severe physical or mental health issues that may affect the learning process.
* Have language comprehension barriers or cognitive impairments, making it difficult to complete learning tasks.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2024-10-20 (Actual); Primary Completion 2025-07-12 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
structured theoretical exam scores | From enrollment to the end of treatment at 4 weeks
  Structured Theoretical Exam Scores - Immediate and One-Month Follow-Up:
  This outcome measures the effectiveness of teaching hypertension management. Students take a structured theoretical exam immediately after the training and again one month later to assess knowledge retention. The exam covers hypertension pathophysiology, risk factors, diagnostics, and treatments. Scores range from 0 to 100, with higher scores indicating better knowledge acquisition and retention.
Clinical Case Test Scores on Hypertension | From enrollment to the end of treatment at 4 weeks
  Clinical Case Test Scores on Hypertension - Immediate and One-Month Follow-Up:This outcome measures how well students apply theoretical knowledge to practical clinical scenarios. Tests are administered immediately after training and one month later, involving clinical simulations where students diagnose hypertension and develop treatment plans. Scores range from 0 to 100, with higher scores indicating better clinical reasoning and application of knowledge.

SECONDARY OUTCOMES:
Mood Elevation Scale | From enrollment to the end of treatment at 4 weeks
  This outcome measures the intensity of emotions felt by students during learning. Participants rate statements on a Likert scale from 1 to 5, where 1 represents "not felt at all" and 5 represents "felt very intensely". Higher scores indicate a stronger emotional response to the learning experience.
Cognitive Load Index (CLI) | From enrollment to the end of treatment at 4 weeks
  This outcome assesses the cognitive load experienced by students during learning. Participants rate statements on a Likert scale from 1 to 5, where 1 represents "strongly disagree" and 5 represents "strongly agree". Higher scores indicate a higher perceived cognitive load during learning.
Teaching Satisfaction Assessment | From enrollment to the end of treatment at 4 weeks
  This outcome evaluates student satisfaction with the teaching methods. Participants rate their experience on a Likert scale from 1 to 5, where 1 represents "strongly disagree" and 5 represents "strongly agree". Higher scores indicate greater satisfaction with the teaching method.
Technology Acceptance Model | From enrollment to the end of treatment at 4 weeks
  This outcome assesses students' acceptance of the GPT system. The questionnaire uses a Likert scale from 1 to 5, where 1 represents "strongly disagree" and 5 represents "strongly agree". Higher scores indicate greater acceptance, usability, and satisfaction with the GPT system.

CONTACTS AND LOCATIONS:
Overall Officials: xianrui luo, Study Chair — The Second Hospital of Anhui Medical University
Locations (1):
- 678 Furong Road, Economic Development Zone, Hefei City, Anhui Province, China, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No